CLINICAL TRIAL: NCT03785457
Title: Immediate Effect Of Standing Trunk Extension Postures On Spinal Height And Clinical Outcome Measures In Low Back Pain: A Randomized Clinical Trial
Brief Title: Standing Trunk Extension and Spinal Height in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L19-024
Record Dates: First submitted 2018-12-12; First posted 2018-12-24 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Extension; Posture; Physical Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The primary investigator will be blinded to the measurements of spinal height using stadiometry, and to the group assignment of each participant (sustained versus repetitive extension postures)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive Trunk Extension (Experimental): Participants with low back pain will be asked to perform standing repetitive trunk extension at a rate of 10 per 45 seconds, repeated five times with 15-second rest breaks
  Interventions: Other: Repetitive Trunk Extension
- Sustained Trunk Extension (Experimental): Participants with low back pain will be asked to perform standing sustained trunk extension for 5 x 45 seconds with 15-second rest breaks
  Interventions: Other: Sustained Trunk Extension

INTERVENTIONS:
Other: Repetitive Trunk Extension — Subjects will be asked to perform standing repetitive trunk extension at a rate of 10 per 45 seconds (Figure 2), repeated five times with 15-second rest breaks.
  Arms: Repetitive Trunk Extension
Other: Sustained Trunk Extension — Subjects will be asked to perform standing sustained trunk extension for 5 x 45 seconds with 15-second rest breaks.
  Arms: Sustained Trunk Extension

SUMMARY:
Background: Standing trunk extension postures have been used for many years as a mechanical approach to low back pain (LBP), sometimes directed by therapeutic intervention, sometimes subconsciously performed by patientsto relieve LBP. However, no study to date has investigated the effect of standing trunk extension postures on spinal height and clinical outcome measures.

Objective: The purpose of this study will be to evaluate in subjects with LBP following a period of trunk loading, how spinal height and/or pain, symptoms' centralization, and function outcome measures respond to:(1) standing repetitive trunk extension posture; and (2) standing sustained trunk extension posture. Lumbar range of motion (ROM) achieved during these two trunk extension postures will be compared to spinal height and outcome measures.

Methods:A pre-test, post-test comparison group design (randomized clinical trial) will be used to determine how spinal height changes in response to sustained and repetitive standing trunk extension after a period of spinal loading. The study will evaluate the effects of sustained and repetitive trunk extension in standing on spinal height, pain, symptoms' centralization and function.

Statistical Analysis: A mixed ANOVA will be used to statistically identify significant interactions and main effects for spinal height, pain and functionoutcome measures. Post-hoc pairwise comparisons will be used to locate significant differences between the different conditions. Significance will be set at α = 0.05. The Kruskal-Wallis 1-factor ANOVA for difference scores will used to determine changes of intensity and location of symptoms following sustained versus repetitive standing trunk extension. Spearman Rank correlation will be used to evaluate the relationship between spinal height changes and changes of pain and location of symptoms for each group.

DETAILED DESCRIPTION:
Standing trunk extension postures have been used for many years as a mechanical approach to low back pain (LBP), sometimes directed by therapeutic intervention, sometimes subconsciously performed by patients to relieve LBP. However, no study to date has investigated the effects of standing extension postures on spinal height, pain, centralization and function. Therefore, the purposes of this study will be to evaluate in a sample of LBP patients the effect of standing trunk extension, both sustained and repetitive, following a period of spinal loading, on (1) spinal height; (2) pain; (3) symptoms centralization and (4) functional measures.

Research Design(s) A pre-test, post-test comparison group design (randomized clinical trial) will be used to determine how spinal height changes in response to sustained and repetitive standing trunk extension after a period of spinal loading. The study will use a 2 (between subjects - type of trunk extension: sustained vs. repetitive) x 3 (within subjects - time: before vs. after vs. 2 weeks after) mixed design to evaluate the effects of sustained and repetitive trunk extension in standing on spinal height, pain, centralization and function outcome measures.

Subjects / Specimens Systematic consecutive sampling of up to 100 subjects with LBP (40 subjects completing both days of data collection) attending "Sports medicine and Physical therapy clinic" in Fredericksburg (Texas) as patients or for the purpose of health and wellness will be recruited. Flyers will also be posted at physician offices and the general Fredericksburg community and surrounding areas to inform subjects about the study.

Testing Sequence Subjects will be asked to attend two physical therapy sessions over approximately a 60-minute period each to complete the study.

SESSION 1

Participants will complete a pre-screening questionnaire regarding inclusion. Each subject will watch an audio-visual power point presentation explaining the study, test procedures and describing the interventions (standing repetitive trunk extension and standing sustained trunk extension). Written informed consent will be obtained. To determine directional preference, the investigator (JH) will use the guidelines set forth in the directional preference definition and based off of standards set forth in randomized clinical trials. Directional preference has been defined as either (1) a specific direction of trunk movement or posture noted during the physical examination or (2) a specific easing factor reported by the patient during the subjective history that alleviates or decreases the patient's pain, with or without the pain having changed location and/or increased the patient's lumbar range of motion. A questionnaire including pertinent medical history will be completed. Subjects will complete (1) a Numerical Pain Rating Scale (NPRS) to rate their current, minimum, maximum and average LBP over the last two days as well as paresthesia signs/symptoms intensity; (2) Body Diagram for indicating location of symptoms; (3) Modified Oswestry low back pain questionnaire; (4) Fear Avoidance Belief Questionnaire. A researcher will record subject's height and weight.

If the subject meets criteria for inclusion in the study, the subject will complete a familiarization procedure to determine the consistency to reposition themselves in the stadiometer. Subjects able to reposition themselves in the stadiometer with a SD of 1.3mm or less for five consecutive measurements will be included in the study. The digital display will be covered to blind the researcher performing the measurements. The data will be automatically recorded by the stadiometer and manually downloaded to a laptop computer.

At the beginning of data collection, a randomization plan generator (http://www.randomization.com ) will assign each subject to one of two interventions: (1) standing repetitive trunk extension at a rate of 10 per 45 seconds, repeated five times with 15-second rest breaks; or (2) standing sustained trunk extension for 5 x 45 seconds with 15-second rest breaks. Each subject will complete one intervention. The intervention number assigned will be recorded by the subject next to their name to allow blinding of the investigator as to which intervention the subject is assigned to. The subject will undergo the test sequence after a 10-minute period of trunk unloading in a supine posture to ensure spinal height is normalized, head in neutral posture, knees supported over a small bolster pillow, hands placed on the abdomen. The subject will reposition on the stadiometer and spinal height will be measured after a relaxed exhalation. The subject then will undergo a five-minute period of loaded upright sitting with a 4.5kg bag secured on each shoulder and spinal height will be measured (Measurement 2). As continued spinal height reduction has been demonstrated following loaded sitting, the subject will undergo an additional five minutes sitting without load and spinal height will be measured (Measurement 3). Inclinometers will be used to take an initial measure of each subject trunk extension prior to intervention. The subject will then undergo one intervention for 5 minutes as previously described, according to the randomization assignment. In order to determine how sustained and repetitive interventions related in terms of change in spinal height, the time to perform the sustained lumbar posture matches the time necessary to perform the repetitive lumbar extension postures.

The subject will reposition on the stadiometer and spinal height will be measured (Measurement 4). Trunk extension will be measured to determine the strength of correlations between the degree of trunk extension during standing trunk extension posture and spinal height, pain and centralization testing outcomes changes. The subject will score their low back and lower extremity symptoms using NPRS, and map their pain on a body pain diagram prior to intervention, immediately after and 2-week following the intervention to determine pain rating and centralization of symptoms. The principal investigator will apply a numeric overlay template to the patient's body diagrams to document the most distal pain location scores between 1 and 6. Higher score will indicate a more distal symptoms' location.

Home instructions Subjects will be instructed to continue to use their medications, including medications aimed at decreasing their pain, as prescribed by their primary healthcare provider and not to change them during the follow-up two-week period. A sheet including home exercise instructions will be provided to each patient. Instructions will include repetitive or sustained trunk extension based on random group assignment, performed approximately 5 times per day. Each subject will complete a sheet recording home exercise compliance upon arrival in session 2.

SESSION 2

Subjects will complete: (1) a NPRS to rate their current, minimum, maximum and average LBP over the last two days as well as paresthesia signs/symptoms intensity; (2) Body Diagram for indicating location of symptoms; (3) Modified Oswestry low back pain questionnaire; (4) Fear Avoidance Belief Questionnaire. Each subject will then complete a familiarization procedure to determine the consistency to reposition themselves in the stadiometer as described in session 1. The subject will undergo a 10-minute period of trunk unloading in a supine posture to ensure spinal height is normalized as described in session 1. The subject will reposition on the stadiometer and spinal height will be measured after a relaxed exhalation (Measurement 1). The subject then will undergo a five-minute period of loaded upright sitting with a 4.5kg bag secured on each shoulder and spinal height will be measured. The subject will then undergo an additional five minutes sitting without load and spinal height will be measured (Measurement 3). Inclinometers will be used to take an initial measure of each subject trunk extension prior to intervention. The subject will then undergo the same intervention as in session 1 for 5 minutes as previously described (standing repetitive trunk extension or standing sustained trunk extension). The subject will reposition on the stadiometer and spinal height will be measured (Measurement 4). Trunk extension will be measured to determine the strength of correlations between the degree of trunk extension during standing trunk extension posture and spinal height, pain and centralization testing outcomes changes. The subjects will then score their low back and lower extremity symptoms using NPRS, and map their pain on a body pain diagram.

Investigator Blinding Two investigators will be involved with data collection and will carry out inclinometer measurements of lumbar and sacral posture, supervised positioning in the stadiometer and stadiometric measurements. The measuring investigator will be blinded to the intervention (each subject will receive a hidden random number and will perform independently the intervention in a treatment room) and the stadiometric measurements during the experiment. He will also be responsible for assigning subjects to their initial groups, supervising the subjects' positioning in the different standing postures and confirming that a stadiometer reading is recorded on an Excel spreadsheet.

Subjects Charges There will be no charge for the two physical therapy sessions, including examination and intervention. Following the two intervention sessions, subjects referred by primary care providers (physicians, chiropractors, nurse practitioners, physician assistants) to physical therapy for LBP will have the choice to receive standard care and be charged for physical therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to come twice to the clinic for approximately 60 minutes each
* Subjects with LBP and directional preference in back extension
* Age 18-80
* Ability to stand for 5 minutes
* Ability to sit for 10 minutes
* Low back pain on Numerical Pain Rating scale (NPRS) of at least 2/10 and less or equal to 9/10

Exclusion Criteria:

* Pregnancy by subject report
* history of back surgery or spinal fractures within the last six months
* history of spinal fusion or physician's diagnosis of spinal instability
* current history of acute systemic infection, active inflammatory disease, or malignancy
* subjects engaged in legal/compensation claims for their back symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Spinal Height (Stadiometry) | Before intervention at first visit
  Spinal height of subjects measured in stadiometer (mm) from 100 to 2000 mm.
Spinal Height (Stadiometry) | Immediately after intervention at first visit
  Spinal height of subjects measured in stadiometer (mm) from 100 to 2000 mm. Height will be compared to height at initial measure. Greater height than at initial measure will indicate height gain.
Spinal Height (Stadiometry) | 2-week following initial visit
  Spinal height of subjects measured in stadiometer (mm) from 100 to 2000 mm. Height will be compared to height at initial measure. Greater height than at initial measure will indicate height gain.

SECONDARY OUTCOMES:
Lumbar Extension range of motion (Inclinometer) | Before intervention at first visit
  Lumbar extension range of motion measured using bubble inclinometers (degrees) from 0 to 180 degrees. Greater numbers indicate greater trunk extension range of motion.
Lumbar Extension range of motion (Inclinometer) | Immediately after intervention at first visit
  Lumbar extension range of motion measured using bubble inclinometers (degrees) from 0 to 180 degrees. Greater numbers indicate greater trunk extension range of motion.
Lumbar Extension range of motion (Inclinometer) | 2-week following initial visit
  Lumbar extension range of motion measured using bubble inclinometers (degrees) from 0 to 180 degrees. Greater numbers indicate greater trunk extension range of motion.
Pain (Numerical pain rating scale - NPRS) | Before intervention at first visit
  Pain (Numerical Pain Rating Scale - NPRS) from 0 (no pain) to 10 (most severe pain requiring emergency room consultation)
Pain (Numerical pain rating scale - NPRS) | After intervention at first visit
  Pain (Numerical Pain Rating Scale - NPRS) from 0 (no pain) to 10 (most severe pain requiring emergency room consultation)
Pain (Numerical pain rating scale - NPRS) | 2-week following initial visit
  Pain (Numerical Pain Rating Scale - NPRS) from 0 (no pain) to 10 (most severe pain requiring emergency room consultation)
Centralization (Dallas Pain Diagram) | Before intervention at first visit
  Centralization of symptoms will be assessed using Dallas Pain diagram. A numeric overlay template will be applied to the patient's body diagram to document the most distal pain location scores between 1 and 6. Higher score will indicate a more distal symptoms' location.
Centralization (Dallas Pain Diagram) | After intervention at first visit
  Centralization of symptoms will be assessed using Dallas Pain diagram. A numeric overlay template will be applied to the patient's body diagram to document the most distal pain location scores between 1 and 6. Higher score will indicate a more distal symptoms' location.
Centralization (Dallas Pain Diagram) | 2-week following initial visit
  Centralization of symptoms will be assessed using Dallas Pain diagram. A numeric overlay template will be applied to the patient's body diagram to document the most distal pain location scores between 1 and 6. Higher score will indicate a more distal symptoms' location.
Modified Oswestry low back pain questionnaire | Before intervention at first visit
  The questionnaire measures how well patient function in life with scale from 0 (normal-no disability) to 100 (crippled with severe disability).
Modified Oswestry low back pain questionnaire | 2-week following initial visit
  The questionnaire measures how well patient function in life with scale from 0 (normal-no disability) to 100 (crippled with severe disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Medicine & Physical Therapy, Fredericksburg, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03785457/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT03785457/ICF_001.pdf